CLINICAL TRIAL: NCT06959589
Title: An Open-label, Multicenter, Single-arm Phase II Clinical Study Evaluating the Efficacy and Safety of IBI351, Cetuximab β Combined With FOLFIRI as First-line /IBI351, Cetuximab β as Second-line in the Treatment of KRAS G12C-mutated Metastatic Colorectal Cancer
Brief Title: The Efficacy and Safety of IBI351, Cetuximab β Combined With FOLFIRI as First-line /IBI351, Cetuximab β as Second-line in the Treatment of KRAS G12C-mutated Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1461
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer Metastatic; KRAS G12C Mutation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI351, cetuximab β+FOLFIRI as first-line treatment/ IBI351+cetuximab β as secon-lfor KRAS G12C mCRC (Experimental)
  Interventions: Drug: IBI351, cetuximab β combined with FOLFIRI

INTERVENTIONS:
Drug: IBI351, cetuximab β combined with FOLFIRI — Cohort A - To evaluate the efficacy and safety of IBI351, cetuximab β combined with FOLFIRI as first-line treatment for metastatic colorectal cancer with KRAS G12C mutations; Twenty untreated patients with advanced colorectal cancer with KRAS G12C mutation are proposed to be enrolled and treated with the first-line IBI351+ cetuximab β injection +FOLFIRI regimen. The historical reference is expected to be around 40-50%, and it is expected to increase to around 75%. Therefore, among the 20 patients, if ≥15 patients achieve remission, it is considered that the efficacy of the trial protocol is statistically significant.
  Cohort B - To evaluate the efficacy and safety of BI351 and cetuximab β as second-line treatment for metastatic colorectal cancer with KRAS G12C mutations.
  It is proposed to enrolled 30 patients with advanced colorectal cancer with KRAS G12C mutation who have progressed after first-line treatment, and evaluate IBI351+ cetuximab β injection for second-line treatment. The hi

SUMMARY:
This is an open-label, multicenter, single-arm Phase II clinical study, divided into subgroups A and B:

Cohort A - To evaluate the efficacy and safety of IBI351, cetuximab β combined with FOLFIRI as first-line treatment for metastatic colorectal cancer with KRAS G12C mutations; Twenty untreated patients with advanced colorectal cancer with KRAS G12C mutation are proposed to be enrolled and treated with the first-line IBI351+ cetuximab β injection +FOLFIRI regimen. The historical reference is expected to be around 40-50%, and it is expected to increase to around 75%. Therefore, among the 20 patients, if ≥15 patients achieve remission, it is considered that the efficacy of the trial protocol is statistically significant.

Cohort B - To evaluate the efficacy and safety of BI351 and cetuximab β as second-line treatment for metastatic colorectal cancer with KRAS G12C mutations.

It is proposed to enrolled 30 patients with advanced colorectal cancer with KRAS G12C mutation who have progressed after first-line treatment, and evaluate IBI351+ cetuximab β injection for second-line treatment. The historical reference is around 25%, and it is expected to increase to around 50%. Therefore, among the 30 patients, if ≥15 patients achieve remission, it is considered that the efficacy of the trial protocol is statistically significant.

Imaging assessment of tumor remission was conducted every 8 weeks until disease progression. The period from the start of treatment to disease progression is defined as PFS. The safety observation indicators include: the incidence and severity of adverse events (AE) and serious adverse events (SAE); Laboratory tests, vital signs, physical examinations, and changes in electrocardiogram (ECG). Record the subsequent tumor treatment and survival follow-up after the progression.

Definition of study conclusion: The study will conclude after the last subject has been treated for 2 years or has completed the treatment (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

The following conditions must be met:

On the day of signing the informed consent form, the age should be ≥18 years old (18-75 years old, including 18 and 75 years old).

2. The patient must have histologically and/or cytologically confirmed metastatic colorectal cancer (stage IV) 3. There is a written test report proving the presence of KRASG12C mutation: PCR method or NGS method detection clearly indicates KRASG12C mutation 4. Cohort A: Untreated advanced metastatic colorectal cancer; Cohort B: Advanced metastatic colorectal cancer with disease progression after first-line standard chemotherapy (FOLFOX,FOLFIRI,XELOX, FOLFOXIRI± targeted therapy) 5. There are measurable lesions according to the Recist 1.1 standard 6.ECOG PS 0-1 7. Weight ≥40Kg 8. Cardiac function test: Left ventricular ejection fraction (LVEF) ≥50%(echocardiography) 9. Life expectancy >3 months 10. Have sufficient organ functions, including:

* There is sufficient hematopoietic function, that is, the absolute neutrophil count (A NC) ≥1.5×109/L, platelet count ≥75×109/L, and hemoglobin ≥9g/d L. Blood transfusion or treatment with granulocyte colony-stimulating factor, thrombopoietin, erythropoietin, etc. shall not be received within 14 days before the blood routine test.
* Have sufficient liver function, namely total bilirubin (TBIL) < 1.5× upper limit of normal value (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (A LT) < 2.5×ULN; If one has Gilbert syndrome, the total bilirubin is less than 2×ULN. If it is liver metastasis of the tumor, the AST and ALT should be less than 5.0×ULN. If direct bilirubin (DBIL) indicates extrahepatic obstruction, TBIL < 3.0×ULN is allowed.
* Have sufficient renal function, that is, creatinine (Cr) ≤1.5×ULN, or when Cr > 1.5×ULN, the creatinine clearance rate (CrCl) calculated using the Cockcroft-Gault formula (see Appendix 5) ≥50 mL/min. Urine protein/creatinine ratio < 1 (or urine analysis < 1+ or 24-hour urine protein < 1g/24 h)
* It has sufficient coagulation function, that is, prothrombin time (PT) and activated partial thromboplastin time (APTT) < 1.5×ULN, and the international normalized ratio (INR) < 1.5 or is within the target range of anticoagulant therapy 11. The toxic reactions of previous anti-tumor treatments need to be restored to the baseline level (except for the residual alopecia effect) or ≤ grade 1 before enrollment (neurotoxicity is acceptable ≤ grade 2). Immune-related Adverse Events (irAE) related to endocrine caused by previous immunotherapy, such as immune-related hypothyroidism that is controlled stably and asymptomatic after treatment, still require stable doses of hormone replacement or physiological doses of corticosteroids for treatment. After the researcher assesses that it does not affect the administration of the study drug and conducts a safety assessment, they can be enrolled 12. Have the ability to take oral medication 13. Fertile female or male subjects must agree to adopt effective contraceptive methods from the date of signing the informed consent form until 30 days after the last administration of IBI351 or 60 days after the last administration of cetuximab. The blood pregnancy test results of fertile female subjects within 7 days (inclusive) before administration should be negative 14. Understand and sign the informed consent form The researchers judged that the subjects could communicate well, be followed up on schedule, and complete the study in accordance with the provisions of the protocol-

Exclusion Criteria:

If any of the following criteria is met, the study must be excluded:

1. Inability to comply with the research protocol or research procedures.
2. dMMR or MSI-H type colorectal cancer.
3. Those who have been confirmed to be allergic to IBI 351, cetuximab β injection and/or its excipients.
4. Have obvious cardiovascular system diseases, such as:

   * Within 6 months, there have been clear cardiovascular abnormal events, such as myocardial infarction, angina pectoris, heart failure, severe arrhythmia, or angioplasty, vascular stent implantation, coronary artery bypass surgery, etc.
   * Clinically significant QT/QTcF interval prolongation (QTcF > 470ms for females or QTcF > 450ms for males).
5. Researchers identify patients with unstable brain metastases. For patients with brain metastases unintentionally detected during the screening process, if they do not cause clinical symptoms and do not require therapeutic intervention, they can be allowed to be enrolled. If the researchers determine that the brain metastasis is stably controlled, the hormone dose is used stably, and the prednisone dose is ≤10mg/d (if other steroid drugs are used, it is the corresponding equivalent dose), enrollment can be allowed.
6. There are significant digestive tract diseases, such as intractable hiccups, nausea, vomiting, severe digestive tract ulcers, liver cirrhosis, active gastrointestinal bleeding, or other diseases that affect the swallowing of tablets or significantly affect the absorption of oral medications;
7. There are major acute or chronic infections, including:

   Active infections that require systemic treatment;
   * Positive human immunodeficiency virus antibody (HIV-Ab) at the baseline period;
   * Active hepatitis B virus infection (positive for hepatitis B surface antigen HBsAg and positive for HBV-D NA); HBsAg was negative and HBcAb was positive. Further examination of HBV-DNA levels is required. If HBV-DNA is positive, the patient will be excluded from the group.
   * Active hepatitis C virus infection (positive hepatitis C antibody HCV-Ab and positive HCV-RNA);
   * Active pulmonary tuberculosis
8. Accompanied by pleural and peritoneal effusion or pericardial effusion that requires repeated drainage or has obvious symptoms.
9. Accompanied by other poorly controlled systemic diseases, such as hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg) that remains uncontrolled even with standardized treatment, diabetes, etc.
10. Within 2 years prior to entering the study, the patient had other malignant tumors, excluding appropriately treated cervical carcinoma in situ, focal cutaneous squamous cell carcinoma, basal cell carcinoma, untreated prostate cancer, ductal carcinoma in situ of the breast, and superficial non-muscular-invasive urothelial carcinoma.
11. Previously received treatment with KRAS G12C inhibitors.
12. Had received therapeutic or palliative radiotherapy within 14 days prior to the administration of this study.
13. Have received other anti-tumor treatments such as chemotherapy, targeted therapy, endocrine therapy, immunotherapy, other investigational drugs or investigational devices within 28 days before administration in this study or within 5 half-lives (whichever is shorter), excluding maintenance endocrine therapy. The patient received treatment with traditional Chinese patent medicines with definite anti-tumor effects within 7 days before the administration of this study.
14. Surgical operations (excluding puncture biopsy) that may affect the administration or evaluation of this study have been performed within 28 days prior to inclusion in this study.
15. Have received strong suppressor or strong inducer of CYP3A4 or P-gp (see Appendix 3) within 14 days before administration in this study or within 5 half-lives of the drug (depending on the longer period), or have taken traditional Chinese medicine within 7 days before administration in this study.

    Those who received known CYP2D6, CYP3A4, P-gp and bCRP-sensitive substrates within 14 days before administration in this study or within 5 half-lives of the drug (whichever is longer), and the therapeutic window of this substrate was relatively narrow, unless enrolled with the unanimous consent of the investigator and sponsor.
16. Pregnant or lactating women. Other circumstances where the researchers consider it unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
ORR | From enrollment to the end of treatment at 8 weeks
  Objective response rate (ORR) : It refers to the proportion of patients whose tumors shrink to a certain extent and remain so for a certain period of time

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided